CLINICAL TRIAL: NCT04219995
Title: Pilot Randomized, Placebo-Controlled Trial to Evaluate The Effect of Oral Pulsed Methylprednisolone on Seizure Frequency in Pediatric Patients With Idiopathic Intractable Convulsive Epilepsy
Brief Title: Pilot Trial to Evaluate The Effect of Oral Methylprednisolone on Seizure Frequency in Children With Epilepsy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB# 19-179
Record Dates: First submitted 2020-01-02; First posted 2020-01-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Intractable Epilepsy; Convulsive Seizures
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional start (Experimental): Patients who randomize to the interventional start arm will receive the study drug, methylprednisolone sodium succinate, in the first month of the study, followed by placebo in the cross-over phase of the study.
  Interventions: Drug: methylprednisolone sodium succinate; Other: Placebo
- Placebo start (Placebo Comparator): Patients who randomize to the placebo start arm will receive placebo in the first month of the study, followed by the study drug, methylprednisolone sodium succinate, in the cross-over phase of the study.
  Interventions: Drug: methylprednisolone sodium succinate; Other: Placebo

INTERVENTIONS:
Drug: methylprednisolone sodium succinate — Methylprednisolone sodium succinate will be re-constituted in simple syrup in a concentration of 80mg/mL and will be administered orally at 20mg/kg (max 1000mg) for days 1, 2, and 3 of the intervention phase of the study.
Other: Placebo — The placebo used in this study will be simple syrup.

SUMMARY:
Although corticosteroids have been shown to be beneficial anecdotally for refractory epilepsy, the effects of corticosteroids on pediatric epilepsy have primarily been studied retrospectively amongst a heterogeneous patient population. The objective of this prospective cross-over study is to determine the effect of oral steroids on convulsive seizure frequency and evaluate the tolerability of pulsed oral steroids. Participants will be prospectively enrolled from pediatric neurology clinic at Children's Hospital of New Orleans, and baseline seizure frequency will be assessed. Participants will then be randomized to receive either the study drug, methylprednisolone, or placebo during the first month, followed by a one-month wash-out period. During the third month of the study, participants will enter the cross-over phase of the study where those who received methylprednisolone will receive placebo, and those who received placebo will receive methylprednisolone. The primary outcome will be the percentage of patients with 50% or more reduction in seizure frequency following one course of oral methylprednisolone. frequency following 1 course of oral methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 2 -18 years of age
2. Patients who have at least 4 convulsive (generalized tonic or tonic-clonic) seizures per month on 2 or more anti-epileptic drugs (AEDs) at therapeutic doses

   a. Epilepsy diagnosed by historical clinical evidence
3. Family's ability to understand and willingness to sign a written informed consent document for patients under 18.
4. Willingness to complete seizure diary for duration of study
5. Willingness to present to all study visits

Exclusion Criteria:

1. Patients with history of the following diagnoses:

   1. Traumatic brain injury
   2. Tuberous sclerosis
   3. Sturge Weber
   4. Cortical dysplasia
2. Patients with known hereditary degenerative diseases as follows:

   1. Adrenoleukodystrophy
   2. Neuronal ceroid lipofuscinosis
   3. Leigh Syndrome
   4. Myoclonic epilepsy with ragged red fibers (MERRF)
   5. Rett Syndrome
3. Patients with the following epilepsy syndromes

   1. Infantile spasms
   2. West Syndrome
   3. Progressive myoclonic epilepsy
   4. Dravet syndrome
   5. Doose syndrome
   6. Ohtahara syndrome
   7. Rasmussen's encephalitis
4. Patients with the following metabolic disorders

   1. Phenylketonuria
   2. Maple syrup urine disease
   3. Organic acidemias
   4. Galactosemia
   5. Peroxismal disorders (e.g. Zellwegers)
   6. Lysosomal disorders
   7. Urea cycle disorders
5. Patients with history of immunodeficiency
6. Patients with the following infections

   1. HIV/AIDS
   2. Active or latent TB
   3. Active or suspected bacterial infection
   4. Active, latent or suspected fungemia
   5. Active or suspected parasitic infection
7. Patients with history of malignancy
8. Patients with history of or active myopathy
9. Patients with degenerative neuromuscular disorders
10. Patients with history of hypersensitivity or allergic reactions to corticosteroids
11. Patients with history of psychosis
12. Patients with diabetes mellitus
13. Pregnancy
14. Any underlying predisposition to gastrointestinal bleeding (peptic ulcer disease, gastritis, colitis)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | The number of seizures per month will be assessed at 1 month (following placebo/intervention), 2 months (following wash-out), and 3 months (following cross-over phase of placebo/intervention). Change compared to baseline will be calculated.
  The percentage of patients with 50% or more reduction in seizure frequency.

SECONDARY OUTCOMES:
Seizure freedom | The number of seizures per month will be assessed at 1 month (following placebo/intervention), 2 months (following wash-out period), and 3 months (following cross-over phase of placebo/intervention).
  The percentage of participants who become seizure free over 1 month
Adverse events | Adverse events will be recorded at 1 month (following placebo/intervention), 2 months (following wash-out period), and 3 months (following cross-over phase of placebo/intervention).
  Percentage of participants who reports adverse events and the severity of the adverse events.
Drop out percentage | The number of participants who drop out will be counted and recorded at 1 month (following placebo/intervention), 2 months (following wash-out period), and 3 months (following cross-over phase of placebo/intervention).
  Percentage of participants who drop out of the study due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Toler, MD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- Children's Hospital of New Orleans, New Orleans, Louisiana, United States